CLINICAL TRIAL: NCT02402023
Title: Novel Treatment to Enhance Smoking Cessation Before Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1407014258; R21CA181569 (NIH)
Record Dates: First submitted 2014-11-17; First posted 2015-03-30 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (SC) (Active Comparator): Patients in the SC arm will receive 4 counseling sessions and nicotine patches as part of typical cessation measures delivered to patients.
  Interventions: Behavioral: Standard of Care (SC)
- Contingency Management (CM) (Experimental): Patients in the CM arm will receive monetary payment contingent on smoking abstinence (in addition to SC: 4 counseling sessions and nicotine patches).
  Interventions: Behavioral: Contingency Management (CM); Behavioral: Standard of Care (SC)

INTERVENTIONS:
Behavioral: Contingency Management (CM) — CM is standard care plus monetary payment delivered contingent on abstinence.
  Arms: Contingency Management (CM)
Behavioral: Standard of Care (SC) — Standard of care consists of smoking cessation counseling sessions and nicotine patches.

SUMMARY:
The purpose of this clinical trial is to determine the feasibility and efficacy of an intervention designed to increase rates of tobacco abstinence for cancer patients before their cancer surgery.

DETAILED DESCRIPTION:
The investigators are proposing a developmental interdisciplinary pilot study to determine the feasibility and efficacy of an intervention designed to increase rates of tobacco abstinence for cancer patients before their cancer surgery. This study (a follow up to smaller pilot studies) will serve as a means to further develop a treatment protocol and to generate an accurate effect size for a full scale trial. The present study will constitute a development clinical trial with a primary aim of developing an effect size for smoking cessation at the time of surgery (7-day point prevalence abstinence), and a secondary aim of creating an effect size for long-term abstinence at 3 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 or older
2. smoking ≥ 1 cigarettes per day
3. CO > 6 ppm
4. diagnosed with or suspicion of any type of operable thoracic, head and neck, breast, or gynecologic cancer
5. agreement on a 2-5-week pre-surgical tobacco intervention by both patient and surgeon, and 6) residence within reasonable driving distance to New Haven.

Exclusion Criteria:

1. unstable psychiatric conditions such as suicidal ideation, acute psychosis, severe alcohol dependence, or dementia
2. unstable medical conditions that have not been well controlled (e.g., acute infection requiring hospitalization) for the past 30 days
3. pregnant or breastfeeding women
4. those with limited decision making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Pre Surgery Smoking Abstinence | Day of Surgery
  Participants will be classified as succeeded or failed in cessation based on a definition of 1 week of abstinence from cigarettes leading up to the day of their surgery based on self-report and confirmed with biochemical verification (CO≤6ppm). For participants who are classified as abstinent, a chi-square will be computed comparing whether treatment with CM is superior to SC in producing a higher probability of abstinence. These data will be used to compute an effect size, Cohen's w, for smoking cessation.

SECONDARY OUTCOMES:
Post Surgery Smoking Abstinence | 3 months
  Participants will be classified 3 months post surgical procedure as succeeded or failed in cessation based on self-report and confirmed with biochemical verification (CO≤6ppm) in the 7 days prior to the 3-month follow-up. For participants who are classified as abstinent, a chi-square will be computed comparing whether treatment with CM is superior to SC in producing a higher probability of abstinence.

OTHER OUTCOMES:
Continuous Smoking Abstinence | 3 months
  This exploratory aim is to assess the continuous days of abstinence 3 months post surgical procedure. It will be calculated from the Timeline Follow Back (TLFB) and will be defined as the number of days from the first date of self-reported abstinence until the first lapse. These data will be collected from intake through the 3-month follow-up. An independent-samples t-test will be used to compare the days of continuous abstinence for those in the CM group versus the SC group.
Perioperative Complications | 3 months
  Wound infections will be assessed (purulent discharge, redness, or serous discharge, including a positive microbial culture or treatment with an antibiotic) 3 months post surgical procedure. This will be recorded from the medical provider interview, along with the duration of the event. The initial dependent measure for this analysis will be the percentage of subjects rated as having wound infections. Instances of respiratory complications (severe coughing, laryngospasm, bronchospasm, recurrent apnea, or pneumonia) will be recorded, along with the duration of the event. The initial dependent measure for this analysis will be the percentage of subjects rated as having respiratory complications. Rates of perioperative complications will be analyzed using a chi-square test comparing CM to SC. Through exploratory step-wise regression modeling of the data, we will attempt to ascertain which variables are important and independent factors with regard to surgical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Toll, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale Cancer Center, New Haven, Connecticut
  - Medical University of South Carolina, Charleston, South Carolina